CLINICAL TRIAL: NCT01720680
Title: Open-label, Prospective Exploratory Study to Assess the Effects of the AlphaCore® Device on Central and Peripheral Airway Dimensions in Patients With COPD
Brief Title: Prospective Exploratory Study to Assess the Effects of the AlphaCore® Device in Patients With COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Wilfried De Backer, Prof. Dr., University Hospital, Antwerp
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PML_DOC_1202
Record Dates: First submitted 2012-10-25; First posted 2012-11-02 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2013-06

CONDITIONS: COPD
Keywords: COPD; Functional Imaging; Patient Reported Outcome (PRO); Lung Function; AlphaCore; Computational Fluid Dynamics
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: Low dose multislice CT thorax — All patients will have 2 low dose multi-slice CT's at visit 2: one CT "pre-dose" and one CT 1 to 3 hours "post-dose".
Device: AlphaCore® device — All patients will receive a stimulation therapy of 90 seconds delivered by the AlphaCore.

SUMMARY:
* Title: Open-label, prospective exploratory study to assess the effects of the AlphaCore® device on central and peripheral airway dimensions in patients with COPD.
* Indication: COPD patients
* Study Design: Open-label, prospective design
* Study Phase: II
* Test treatment duration: 1 day
* Test treatment: AlphaCore® device
* Dosage regimen: 1 session of stimulation during 90 seconds
* Patient number: up to 10 evaluable patients with COPD
* Patient age: ≥ 18 years
* Sex: male or female
* Primary objective: The evaluation of the effect of the AlphaCore® device on central and peripheral airway dimensions with Computational Fluid Dynamics (CFD).
* Secondary objectives: The assessment of the effect of the AlphaCore® device on lung function (spirometry, diffusion and resistance) and on patient reported outcomes (PRO's).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a documented diagnosis of COPD
* Male or female patients aged ≥18 years
* Patients with a co-operative attitude to be treated with the AlphaCore® device
* Patients should take anti-cholinergics
* Female patient of childbearing potential who confirm to use a contraception method during the study
* Written informed consent obtained

Exclusion Criteria:

* Pregnant or lactating females or females at risk of pregnancy at screening and not willing to use an appropriate contraception method during the study period
* Inability to carry out pulmonary function testing
* Patients with an uncontrolled disease or any condition that might, in the judgement of the investigator, place the patient at undue risk or potentially compromise the results or interpretation of the study
* Patients with an electrical and/or neurostimulator device (e.g. a cardiac pacemaker, a vagal neurostimulator, a defibrillator, a cochlear implant, …)
* Patients with an abscess or other infection or lesion (incl. lymphadenopathy) at the therapy head placement site
* Patients with a compromised cervical anatomy (such as from scaring, infection or suspected carotid artery disease) or a cervical vagotomy
* Patients with a history of carotid endarterectomy or vascular neck surgery on the right side
* Patients with coagulopathy, irregular heart rhythm or that are on pressor medication
* Patients unlikely to comply with the protocol or unable to understand the nature, scope and possible consequences of the study
* Patients who received any investigational new drug within the last 4 weeks prior to the screening visit
* Patients treated with any non-permitted concomitant medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-10; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Changes in functional imaging parameters | At V2 (2 - 14 days after screening) pre and post treatment with the AlphaCore device
  The primary objective of this study is to evaluate the effect of the AlphaCore® on central and peripheral airway dimensions with functional imaging using airway segmentation and computational methods (CFD).

SECONDARY OUTCOMES:
Changes in lung function parameters | At V2 (2 - 14 days after screening) pre and post treatment with the AlphaCore device
  The secondary objectives of this study are to assess the effects after treatment with the AlphaCore® on lung function (spirometry, resistance and diffusion), on COPD Assessment Test (CAT), on Modified Medical Research Council (MMRC), on Saint George's Respiratory Questionnaire (SGRQ) and on health questionnaire EQ-5D-5L.
Changes in patient reports outcomes (PROs) | At V2 before treatment with the AlphaCore device and at follow-up visit (14 days after visit 2)
  The secondary objectives of this study are to assess the effects after treatment with the AlphaCore® on lung function (spirometry, resistance and diffusion), on COPD Assessment Test (CAT), on Modified Medical Research Council (MMRC), on Saint George's Respiratory Questionnaire (SGRQ) and on health questionnaire EQ-5D-5L.

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried De Backer, MD, PhD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- University Hospital Antwerp, Edegem, Antwerp, Belgium